CLINICAL TRIAL: NCT02245659
Title: The Effect of Continuous Positive Airway Pressure (CPAP) Treatment on Glycemic Control in Gestational Diabetes: A Pilot Randomized-Controlled Trial
Brief Title: Effect of CPAP Treatment on Glycemic Control in Gestational Diabetes: A Pilot Randomized-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sushmita Pamidi, Assistant Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RN-326488
Record Dates: First submitted 2014-04-25; First posted 2014-09-19 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy; Sleep-disordered Breathing; Gestational Diabetes
MeSH Terms: conditions — Sleep Apnea Syndromes; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental)
  Interventions: Device: CPAP
- Nasal dilator strip (Other): Control
  Interventions: Other: Nasal dilator strip

INTERVENTIONS:
Device: CPAP — Continuous Positive Airway Pressure
  Arms: CPAP
Other: Nasal dilator strip — Nasal dilator strip to be worn nightly
  Other Names: Breathe-Right Strip
  Arms: Nasal dilator strip

SUMMARY:
Clinical trial on effects of continuous positive airway pressure (CPAP) on glucose levels in pregnant patients with sleep-disordered breathing and gestational diabetes

DETAILED DESCRIPTION:
Gestational diabetes (GDM), defined as glucose intolerance that is first recognized during pregnancy, is associated with adverse maternal and fetal outcomes. Sleep-disordered breathing (SDB) is characterized by breathing pauses during sleep leading to recurrent arousals and intermittent hypoxia. The resulting increases in sympathetic drive, cortisol and inflammation have been shown to lead to glucose dysregulation. In that SDB is prevalent during pregnancy, SDB may represent a novel risk factor for GDM, as suggested by recent observational studies. No interventional studies evaluating the effects of SDB treatment on GDM outcomes have yet been published.

General Objective: To perform a pilot study to assess the feasibility of conducting a randomized-controlled trial using continuous positive airway pressure (CPAP) to evaluate the effects of SDB treatment on maternal-fetal outcomes in GDM.

Primary Aim of Pilot Study: 1) To assess CPAP adherence in pregnant patients with GDM. Secondary Aims: 2) To assess recruitment and retention rates over ~2 months of treatment 3) To assess adequacy of nasal dilator strips as the control intervention 4) To measure maternal glucose levels to determine sample size calculations for a future large-scale multi-site randomized-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥ 18 y referred to the GDM clinic at the McGill University Health Centre
* >20 weeks and <34 weeks gestational age at time of recruitment
* Gestational diabetes
* Sleep-disordered breathing (SDB)

Exclusion Criteria:

* Pre-gestational type 1 or type 2 diabetes
* Multiple pregnancy
* Conception by IVF
* Prior treatment for SDB
* severe medical illness
* Severe SDB (AHI >30) and Epworth Sleepiness Scale >15 or oxygen desaturation index >30 or sustained hypoxia < 80%
* Habitual sleep duration on average less than 5 hours/night (determined by actigraphy)
* Cigarette smoking, alcohol consumption or illicit drug use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Average nightly hours of CPAP use | Up to 8 weeks
  Calculated over the course of pregnancy, with objective measurement from CPAP device download. CPAP will be initiated at time of diagnosis of sleep apnea after GDM diagnosis, and up until delivery of the baby (expected duration of 6-8 weeks)

SECONDARY OUTCOMES:
Recruitment and retention rates in trial | At completion of study (prior to delivery of baby)
Maternal glucose levels | Throughout pregnancy until delivery
  Continuous glucose monitoring and capillary blood glucose checks

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smocot J, Huynh N, Panyarath P, Kimoff RJ, Meltzer S, Drouin-Gagne L, Newbold R, Hebert C, Benedetti A, Arcache JP, Morency AM, Garfield N, Rey E, Pamidi S. Patterns of adherence to continuous positive airway pressure and mandibular advancement splints in pregnant individuals with sleep-disordered breathing. Sleep Breath. 2025 Apr 4;29(2):148. doi: 10.1007/s11325-025-03284-5. PMID 40183988
- [Derived] Pamidi S, Meltzer SJ, Garfield N, Lavigne L, Olha A, Khalyfa A, Benedetti A, Tremblay G, Gagnon R, Rey E, Dasgupta K, Kimoff RJ. A Pilot Randomized-Controlled Trial on the Effect of CPAP Treatment on Glycemic Control in Gestational Diabetes: Study Design and Methods. Front Endocrinol (Lausanne). 2018 Nov 16;9:659. doi: 10.3389/fendo.2018.00659. eCollection 2018. PMID 30505290